CLINICAL TRIAL: NCT02206191
Title: The Primary Care Obesity Network (PCON): Incorporating Principles of Self-regulation of Intake
Acronym: PCON
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Ihuoma Eneli, Director, Center for Healthy Weight and Nutrition; Professor of Pediatrics, The Ohio State University, Nationwide Children's Hospital
Other Study IDs: IRB13-00262; Food Innovation Center (Other Grant/Funding Number: The Ohio State University)
Record Dates: First submitted 2014-07-21; First posted 2014-08-01 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Self-regulation
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mothers of 6-11 year olds

SUMMARY:
In response to the high prevalence rates of childhood obesity in central Ohio, the Center for Healthy Weight and Nutrition (CHWN) established the Primary Care Obesity Network (PCON); a partnership between primary care physicians and Nationwide Children's Hospital's Center for Healthy Weight and Nutrition, a tertiary care obesity center, the first of its kind in Ohio. The overall goal of PCON is to bring an effective and user friendly obesity management program to the community physician's office to prevent and treat the growing number of obese children in the setting of the private office. The predominant nutrition messaging approach to tackling childhood obesity has revolved around the food choices and portion sizes. While this is relevant, an area with significant potential for impact for maintaining optimal growth and a healthy weight for young children is addressing feeding behaviors and self-regulation of intake;. - the "how" of eating. The investigators objective it to investigate whether this self-regulation approach can be employed for an older age group of 6-11 years old.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a 6-11 year old child

Exclusion Criteria:

* Unable to speak and read English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mothers of 6-11 year olds being seen in primary care offices throughout Columbus, OH.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Examining use of disordered self-regulatory feeding behaviors, at survey completion | At survey completion, which will occur about 30 minutes after the survey is administered

CONTACTS AND LOCATIONS:
Overall Officials: ihuoma Eneli, MD, Principal Investigator — Nationwide Childrens Hospital, Columbus, Ohio
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States